CLINICAL TRIAL: NCT06326541
Title: The Effect of Listening to the Holy Quran on Life Findings in Coma Patients Hospitalized in Surgical Intensive Care Unit
Brief Title: The Effect of Listening to the Holy Quran on Vital Signs in Coma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, principal ınvestigator, Bitlis Eren University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: okutan
Record Dates: First submitted 2024-03-06; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Sequelae of; Complications Surgical and Medical Care
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: single group pretest-posttest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- music therapy (Experimental): music therapy
  Interventions: Behavioral: music therapy

INTERVENTIONS:
Behavioral: music therapy — Listening to the Holy Quran.

SUMMARY:
The aim of this study is to examine the effect of the Holy Quran listened to to coma patients on their vital signs.

Does listening to the Holy Quran have a positive effect on the life values of coma patients?

DETAILED DESCRIPTION:
This study aims to examine the effect of listening to the Holy Quran on vital signs (fever, pulse, respiration, systolic-diastolic blood pressure, saturation) in surgical intensive care unit patients. The unique value of this study, unlike other studies, is to examine the positive changes in patients' vital signs by listening to the Holy Quran (Surah Rahman) instead of classical music.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Being a surgical intensive care patient
* Having a Glasgow coma score of 8 points or less

Exclusion Criteria:

* The patient must be under 18 years of age
* Have a Glaskow coma score above 8 points
* Be out of coma during the time the research continues

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure- (mmHg) | 30 minutes
  Vital Signs Values of Patients Before and After Application
diastolic blood pressure- (mmHg) | 30 minutes
  Vital Signs Values of Patients Before and After Application
pulse (number of beats/min) | 30 minutes
  Vital Signs Values of Patients Before and After Application
body temperature (degrees Celsius) | 30 minutes
  Vital Signs Values of Patients Before and After Application
saturation (%-oxygen saturation) | 30 minutes
  Vital Signs Values of Patients Before and After Application

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, Dr., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yorke J, Wallis M, McLean B. Patients' perceptions of pain management after cardiac surgery in an Australian critical care unit. Heart Lung. 2004 Jan-Feb;33(1):33-41. doi: 10.1016/j.hrtlng.2003.09.002. PMID 14983137